CLINICAL TRIAL: NCT05413850
Title: An Open-label, Multicentre, Integrated Phase 1 & 2 Study to Evaluate the Safety, Tolerability, Radiation Dosimetry and Anti-tumour Activity of Lutetium (177Lu) rhPSMA-10.1 Injection in Men With Metastatic Castrate-resistant Prostate Cancer
Brief Title: Anti-tumour Activity of (177Lu) rhPSMA-10.1 Injection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Blue Earth Therapeutics Ltd (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BET-PSMA-121
Record Dates: First submitted 2022-05-20; First posted 2022-06-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; mCRPC; Urogenital Neoplasms; Prostatic Neoplasms; Prostatic Diseases
Keywords: PSMA; mCRPC; Prostate cancer; 177Lu rhPSMA-10.1; 18F-rhPSMA-7.3; BET-PSMA-121; Blue Earth Therapeutics Limited; Radiohybrid; Radiopharmaceuticals
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms; Prostatic Diseases | interventions — Lutetium; Lutetium-177

STUDY DESIGN:
Intervention Model Description: Non Randomized (Phase 1) and Randomized (Phase 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1, Cohort A (Experimental): Subjects with PSMA positive disease will receive 5.55GBq of 177Lu-rhPSMA-10.1 (maximum of 3 cycles).
  Interventions: Drug: Lutetium (177Lu) rhPSMA-10.1 Injection; Diagnostic Test: 18F-rhPSMA-7.3 injection (in phase 1 only)
- Phase 1, Cohort B (Experimental): Subjects with PSMA positive disease will receive 7.4GBq of 177Lu-rhPSMA-10.1 (maximum of 3 cycles).
  Interventions: Drug: Lutetium (177Lu) rhPSMA-10.1 Injection; Diagnostic Test: 18F-rhPSMA-7.3 injection (in phase 1 only)
- Phase 2, Cohort 2A (Experimental): Subjects with PSMA positive disease will receive 2 doses at 10.00 GBq (270 mCi) followed by up to 5 additional doses at 7.40 GBq (200 mCi), all doses administered at 6-weekly intervals.
  Interventions: Drug: Lutetium (177Lu) rhPSMA-10.1 Injection
- Phase 2, Cohort 2B (Experimental): Subjects with PSMA positive disease will receive up to 8 doses at 7.40 GBq (200 mCi). The first 3 doses will be administered at 3-weekly intervals, with the remaining doses being administered at 6-weekly intervals.
  Interventions: Drug: Lutetium (177Lu) rhPSMA-10.1 Injection
- Phase 2, Cohort 2C (optional) (Experimental): If opened, subjects with PSMA positive disease will receive 2 doses at 14.80 GBq (400 mCi) followed by up to 4 additional doses at 7.40 GBq (200 mCi), all doses administered at 6-weekly intervals.
  Interventions: Drug: Lutetium (177Lu) rhPSMA-10.1 Injection

INTERVENTIONS:
Drug: Lutetium (177Lu) rhPSMA-10.1 Injection — Therapeutic cycles of 177Lu-rhPSMA-10.1
  Other Names: 177Lu-rhPSMA-10.1
Diagnostic Test: 18F-rhPSMA-7.3 injection (in phase 1 only) — 18F-rhPSMA-7.3 (in phase 1 only) at an administered activity of 296 MBq (8 mCi) for PET/CT scan to ascertain whether the subject has PSMA-positive disease.
  Other Names: 18F-rhPSMA-7.3 (in phase 1 only)
  Arms: Phase 1, Cohort A; Phase 1, Cohort B

SUMMARY:
To determine the dose, safety, radiation dosimetry and efficacy of 177Lu-rhPSMA-10.1 in participants with PSMA-expressing metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
This is an interventional, open-label, integrated Phase 1 & 2 study to assess the safety, tolerability, radiation dosing regimen and anti-tumour activity of Lutetium (177Lu) rhPSMA-10.1 (IMP) in men with metastatic castrate-resistant prostate cancer (mCRPC). The study will consist of 2 parts: a non-randomised Phase 1 part, with safety, dose-finding, and dosimetry components, and a randomised Phase 2 part, with efficacy and safety assessments, and testing dosing regimens selected following analysis of the safety and dosimetry data in Phase 1. Both phases will include subjects with prostate-specific membrane antigen (PSMA)-positive mCRPC, which has progressed following prior therapy. Phase 1 will include a post-chemotherapy mCRPC cohort of subjects who have experienced disease progression on or after at least 1 novel androgen axis drug (NAAD) (e.g. abiraterone, enzalutamide) and at least 1 course (but no more than 2 courses) of taxane-based chemotherapy. Phase 2 will include subjects who have experienced disease progression on or after at least 1 NAAD (e.g. abiraterone, enzalutamide, apalutamide, darolutamide) but have not received previous taxane-based chemotherapy for the treatment of mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, 18 years of age or older with histologically confirmed adenocarcinoma of the prostate.
2. Serum testosterone levels <50 ng/dL (1.73 nmol/L) after surgical or continued chemical castration.
3. Presence of disease target or non target lesions (per RECIST v1.1) on CT/MRI and/or presence of disease on full body 99mTc bone scan performed within 28 days of screening.
4. Positive disease expression of PSMA as confirmed on PSMA PET/CT scan.
5. At least 4 weeks or 5 half-lives (whichever is longer) elapsed between last anti-cancer treatment administration and the initiation of study treatment (except for Luteinising Hormone-releasing Hormone or GnRH).
6. Resolution of all previous treatment related toxicities to CTCAE version 5.0 grade of ≤1 (except for chemotherapy induced alopecia and grade 2 peripheral neuropathy or grade 2 urinary frequency which are allowed).
7. Prior major surgery must be at least 12 weeks prior to study entry.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 with a life expectancy ≥6 months.
9. Adequate bone marrow reserve and organ function as demonstrated by blood count, and serum biochemistry at baseline.
10. Adequate contraception for patients and their partners.
11. For Phase 1 mCRPC only: Subjects who have experienced disease progression on or after at least 1 NAAD (e.g. abiraterone, enzalutamide) and at least 1 course (but no more than 2 courses) of taxane-based chemotherapy. For Phase 2 mCRPC only: Subjects who have experienced disease progression on or after at least 1 NAAD (e.g. abiraterone, enzalutamide, apalutamide, darolutamide), but have not received previous taxane-based chemotherapy for the treatment of mCRPC.

Exclusion Criteria:

1. Known hypersensitivity to the therapeutic or diagnostic IMP or any of its constituents.
2. Presence of significant PSMA-negative disease on ceCT/MRI scan
3. Diffuse marrow infiltration of disease ('superscan' appearance on full body 99mTc bone scan).
4. Symptomatic spinal cord compression, or clinical or radiological findings that are indicative of impending spinal cord compression.
5. Known history of haematological malignancy.
6. Known history of central nervous system (CNS) metastases.
7. Histological findings consistent with neuroendocrine phenotype of prostate cancer.
8. Known history of other solid malignancy that may reduce life expectancy and/or may interfere with disease assessment.
9. Unresolved urinary tract obstruction defined as radiographic evidence of hydronephrosis with or without ureteric stent/nephrostomy.
10. Any uncontrolled significant medical, psychiatric, or surgical condition or laboratory finding that would pose a risk to subject safety or interfere with study participation or interpretation of individual subject results.
11. Ongoing treatment with bisphosphonates for bone-targeted therapy.
12. Severe urinary incontinence that would preclude safe disposal of radioactive urine.
13. Single kidney or renal transplant or any concomitant nephrotoxic therapy that might put the subject at high risk of renal toxicity during the study in the judgement of the investigator.
14. Clinically significant abnormalities on a single 12 lead electrocardiogram (ECG) at screening.
15. Previously received external beam irradiation to a field that includes more than 30% of the bone marrow or kidneys.
16. Previous treatment with any of the following: PSMA targeted radionuclide therapy, Strontium-89, Samarium-153, Rhenium 186, Rhenium-188, Radium-223, hemi-body irradiation.
17. Subjects with bilateral hip replacements or any significant metallic implants or objects, that may affect image quality and/or dosimetry calculations.
18. Transfusion of blood products for the sole purpose of meeting the eligibility criteria for this clinical study.
19. Participation in other studies involving IMP(s) within 28 days or 5 half-lives (whichever is longer) prior to study entry and/or during study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Incidence of DLTs | 6 weeks post final IMP
  Incidence of DLTs during the DLT observation period.
Phase 1 Frequency and nature of TEAEs | End of study
  Frequency and nature of treatment-emergent adverse events (TEAEs).
Phase 2 Evaluate the efficacy of Lutetium (177Lu) rhPSMA-10.1 Injection | 6 weekly intervals
  The number of subjects with an anti-tumour response defined as ≥50% reduction in PSA level from baseline to the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Blue Earth Therapeutics, Study Director — Blue Earth Therapeutics
Locations (14):
- United States (4):
  - Biogenix Molecular LLC, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Weill Cornell Medicine - New York - Presbyterian Hospital, New York, New York
- Belgium (4):
  - Jules Bordet Institute, Brussels
  - Saint Luc University Hospital, Brussels
  - University Hospital Ghent, Ghent
  - University Hospital Center Sart-Tilman, Liège
- Radboud UMC, Nijmegen, Gelderland, Netherlands
- United Kingdom (5):
  - Bristol Hematology and Oncology Center, Bristol
  - Beatson West of Scotland Cancer Center, Glasgow
  - St Bartholomew's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dierks A, Gable A, Rinscheid A, Wienand G, Pfob CH, Kircher M, Enke JS, Janzen T, Patt M, Trepel M, Weckermann D, Bundschuh RA, Lapa C. First Safety and Efficacy Data with the Radiohybrid 177Lu-rhPSMA-10.1 for the Treatment of Metastatic Prostate Cancer. J Nucl Med. 2024 Mar 1;65(3):432-437. doi: 10.2967/jnumed.123.266741. PMID 38164586
- See also: Sponsor website — http://www.blueearththerapeutics.com